CLINICAL TRIAL: NCT06862869
Title: Real World Clinical Outcomes of Resected ALK-Positive Early Stage NSCLC Patients Treated With Alectinib as Adjuvant Therapy in China: A Multicenter, Prospective Cohort Study
Brief Title: Real World Clinical Outcomes of Resected ALK-Positive Early Stage NSCLC Patients Treated With Alectinib as Adjuvant Therapy
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML45766
Record Dates: First submitted 2025-02-20; First posted 2025-03-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with resected stage II-IIIB ALK-positive NSCLC who have received Alectinib adjuvant therapy will be followed-up for approximately 2.5 years during routine visits at real-world clinical practice settings.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will have received alectinib adjuvant treatment for resected stage II-IIIB ALK-positive NSCLC in routine clinical practice.
  NOTE: No intervention will be provided in this study as the study is observational.

SUMMARY:
This study is a multicenter, prospective, cohort study designed to evaluate the clinical outcomes and characteristics of resected stage II-IIIB anaplastic lymphoma kinase (ALK)-positive non-small-cell lung cancer (NSCLC) adult patients treated with Alectinib as adjuvant therapy in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed stage II-IIIA or selected IIIB (T3N2) NSCLC as per the American Joint Committee on Cancer and International Union Against Cancer (UICC/AJCC), 8th edition
* ALK positive
* Postoperative NSCLC patients who have undergone complete resection
* Had taken Alectinib monotherapy without prior systemic therapy (including other ALK-TKIs or chemotherapy) as adjuvant† therapy for resected stage II-IIIB ALKpositive NSCLC and the time from the first dose to enrollment was no more than 28 days

Exclusion Criteria:

* Patients participating in interventional study of adjuvant treatment
* Pregnant, lactating, or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in China with resected stage II-IIIB ALK-positive NSCLC treated with adjuvant Alectinib according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Real-world disease-free survival (rwDFS) | From baseline to the date of the first documentation of cancer recurrence, as determined by the physician according to local clinical standard of care, or death due to any cause, whichever occurs first (up to approximately 2.5 years)

SECONDARY OUTCOMES:
Duration of alectinib therapy | From start of treatment to the date of treatment discontinuation (up to approximately 2.5 years)
Participant demographics by disease stage and city tier | Up to approximately 2.5 years
Participant clinical characteristics as determined by Eastern Cooperative Oncology Group performance status (ECOG PS) by disease stage and city tier | Up to approximately 2.5 years
Participant clinical characteristics as determined by surgery history by disease stage and city tier | Up to approximately 2.5 years
Emotional and physical functioning as determined by the 36-item short form survey (SF-36) v2 questionnaires | At enrollment, then every approximately 3 months thereafter (up to approximately 2.5 years)
Incidence and severity of adverse events (AEs) | Baseline to withdrawal from study or 28 days after the last dose of alectinib, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- China (35):
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangzhou
  - Huai He Hospital of Henan University, Kaifeng, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Changzhou First People's Hospital, Changzhou
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - Huzhou Central Hospital, Huzhou
  - Jiangmen Central Hospital, Jiangmen
  - Shandong Provincial Hospital, Jinan
  - Lanzhou University Second Hospital, Lanzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo No.2 Hospital, Ningbo
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Liaoning Provincial Cancer Hospital, Shengyang
  - Hebei Medical University Fourth Hospital, Shijiazhuang
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Chest disease hospital of Tianjin City, Tianjin
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Xi'an International Medical Center Hospital, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No